CLINICAL TRIAL: NCT01819402
Title: Effects of Pioglitazone on Visceral Fat Metabolic Activity
Brief Title: Pioglitazone Decreases Visceral Fat Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Nobuhiro Tahara, MD, PhD, Kurume University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIO FAT
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: To Evaluate the Effect of Pioglitazone on Glucose Metabolism of Fat Tissue by Using FDG-PET/CT Imaging
Keywords: visceral fat metabolism; FDG-PET/CT; pioglitazone; glimepiride; adiponectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator: 1 (Active Comparator): up to 30 mg pioglitazone, tablet, orally, once daily
  Interventions: Drug: Pioglitazone vs Glimepiride
- Sham Comparator: 1 (Sham Comparator): up to 4 mg/day glimepiride, tablet, orally, once daily
  Interventions: Drug: Pioglitazone vs Glimepiride

INTERVENTIONS:
Drug: Pioglitazone vs Glimepiride

SUMMARY:
Excess visceral fat is associated with chronic systemic inflammation and cardiovascular complications. Pioglitazone has been reported to variably influence visceral fat volume, but it its effect on metabolic activity of the visceral fat remains uncharacterized. To evaluate the effect of pioglitazone on glucose metabolism of fat tissue by using 18F-fluorodeoxyglucose (FDG)-positron emission tomography (PET) and computed tomography (CT) imaging.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 35 and 85 years
* Subjects with impaired glucose tolerance and type 2 diabetes

Exclusion Criteria:

* Subjects with insulin treatment
* Subjects with uncontrolled diabetes, hypertension, symptomatic coronary artery disease, symptomatic cerebrovascular disease
* Subjects taking more than three antidiabetic medications
* Subjects taking anti-platelet, statins, antidiabetic agents, thiazolidinediones within 8 weeks prior to randomization
* Subjects with cardiac failure (New York Heart Association Class > III) or left ventricular dysfunction (LVEF < 40%)
* Subjects with systemic disorders such as active inflammatory, liver, renal, hematopoietic, and malignant disease

Ages: 35 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Effect of treatment on the nominal change in FDG uptake of fat tissue from baseline after 16 weeks of treatment as measured by FDG-PET/CT imaging. | Baseline and 16 weeks after treatment

SECONDARY OUTCOMES:
Change from baseline in plasma glucose/insulin homeostatic parameters and circulating inflammatory markers | Baseline and 16 weeks after treatment

OTHER OUTCOMES:
All cardiovascular events and all cause death for 5 years | Baseline and 5 years after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kurume University, Kurume, Japan